CLINICAL TRIAL: NCT03864640
Title: Reliability and Validity of Mediterranean Colorectal Cancer Registry
Status: Completed | Type: Observational
Sponsor: Volkan Doğru (Other)
Responsible Party: Sponsor-Investigator, Volkan Doğru, Öğretim Görevlisi Doktor, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: 19920022019
Record Dates: First submitted 2019-02-27; First posted 2019-03-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Registries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer: Patients with colorectal cancer

SUMMARY:
The study will examine the validity and reliability of the Mediterranean Colorectal Cancer Registry. Aspects of the analysis will cover parallel forms reliability, test-retest reliability, split half internal consistency and face validity of the Mediterranean Colorectal Cancer Registry.

DETAILED DESCRIPTION:
Although central cancer registry programs have many benefits (the determination of national cancer incidences, strategic planning of health care systems etc.) data entry in such programs is often collected in restricted variables and physicians participating in the registration process may not be able to interact with each other during the management of their patients. For these reasons, a complete record in national general cancer registries can only be established retrospectively and the direct contribution to patient-specific diagnosis / treatment is limited. On the other hand, local registries have many advantages like easy integration of the data into the hospital electronic systems and multidisciplinary proactive enrollment.

Thus, characteristics of ongoing colorectal cancer registries (Swedish, South Australian, Oregon, Lublin, Ontario etc.) reported previously in the English medical literature are reviewed and an electronic form is tabulated for the Mediterranean Colorectal Cancer Registry. This study will examine the validity and reliability of this registry. Aspects of the analysis will cover construct validity, content validity, parallel forms reliability, test-retest reliability, split half internal consistency and face validity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with colorectal cancer.

Exclusion Criteria:

* Patients reluctant to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patients with colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Construct validity of Mediterranean Colorectal Cancer Registry: answering multiple-choice items | 2 week
  Construct validity will be based on the combination of qualitative and statistical methods in order to develop representative and structured set of multiple-choice items for colorectal cancer registry.
Content validity of Mediterranean Colorectal Cancer Registry: answering multiple-choice items | 2 week
  Content validity will be based on the combination of qualitative and statistical methods in order to develop shortest-possible but well-matched set of multiple-choice items reflecting the subjects being assessed in the colorectal cancer registry. .

SECONDARY OUTCOMES:
Parallel forms reliability of Mediterranean Colorectal Cancer Registry: answering multiple-choice items | 2 week
  Parallel forms reliability will be based on assessments analyzing the extent to which the items answered by different responders correlate with each other within their domain. It will be evaluated by correlation scores or positive predictive values according to the subject being assessed.
Test-retest reliability of Mediterranean Colorectal Cancer Registry: answering multiple-choice items | 2 week
  Test-retest reliability will be based on the reproducibility of the answers to multiple-choice items during a specific time period of stable condition. It will be evaluated by intraclass correlation coefficient or positive predictive values according to the subject being assessed.
Split half internal consistency of Mediterranean Colorectal Cancer Registry: answering multiple-choice items | 2 week
  Split half internal consistency will be based on the comparison of two sets of items inquirying the same subject. It will be evaluated by correlation scores or positive predictive values according to the subject being assessed.
Face validity of Mediterranean Colorectal Cancer Registry: binary scoring of items | 2 week
  Face validity will be based on the scores of respondents indicating their overall positive or negative impression after evaluating each item for every file they registered.
Face validity of Mediterranean Colorectal Cancer Registry: the major reason behind the negative response | 2 week
  For negative responses, respondents will provide further feedback whether the item was ambiguous, confusing, excessively short, excessively long or there was another reason for their negative impression.

CONTACTS AND LOCATIONS:
Overall Officials: Muhittin Yaprak, Study Director — Akdeniz University Hospital
Locations (1):
- Muhittin Yaprak, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided